CLINICAL TRIAL: NCT06485947
Title: Phase Ib Study Combining Dinutuximab Beta With Induction Chemotherapy Regimens in Patients With Newly Diagnosed High-risk Neuroblastoma
Brief Title: Study Combining Dinutuximab Beta With Two Chemotherapy Regimens in Neuroblastoma
Acronym: DBPilot
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: EUSA Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIOPEN-Pilot01.; 2023-509673-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-15; First posted 2024-07-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dinutuximab Beta with chemotherapy treatment called GPOH (Experimental): Dinutuximab Beta will be administered at a fixed daily dose of 10 mg/m2 given as a 24-hour continuous infusion for a scheduled number of days within each treatment cycle of chemotherapy.
  Interventions: Biological: Dinutuximab beta; Drug: chemotherapy treatment called GPOH
- Dinutuximab Beta with chemotherapy treatment called rapid COJEC (Experimental): Dinutuximab Beta will be administered at a fixed daily dose of 10 mg/m2 given as a 24-hour continuous infusion for a scheduled number of days within each treatment cycle of chemotherapy.
  Interventions: Biological: Dinutuximab beta; Drug: chemotherapy treatment called rapid COJEC

INTERVENTIONS:
Biological: Dinutuximab beta — Combination of immunotherapy with standard chemotherapy
  Other Names: Immunotherapy
Drug: chemotherapy treatment called GPOH — chemotherapy treatment called GPOH
  Arms: Dinutuximab Beta with chemotherapy treatment called GPOH
Drug: chemotherapy treatment called rapid COJEC — chemotherapy treatment called rapid COJEC
  Arms: Dinutuximab Beta with chemotherapy treatment called rapid COJEC

SUMMARY:
The goal of this clinical trial is to to assess the dose level of dinutuximab Beta (DB) when combined with 2 different induction chemotherapy regimens (named GPOH or rapid COJEC) in newly diagnosed high-risk neuroblastoma patients. The main question is:

• to assess the safety and tolerability and identifying the recommended phase II dose and/or the maximum tolerable dose of dinutiximab Beta when combined with 2 standard induction chemotherapy regimens

Participants will receive:

* GPOH + dinutuximab beta infusion duration = 10 mg/m2 × 5 days (50 mg/m2/course) in 21-day treatment intervals.
* Rapid COJEC + dinutuximab beta infusion duration = 10 mg/m2 × 3 days (30 mg/m2/course) in 10-day treatment intervals.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, dual-cohort, Phase 1 study of DB combined with each of 2 different induction chemotherapy regimens in 2 cohorts. When the recommended cumulative DB dose level has been defined for each of the chemotherapy regimens, a confirmation cohort of 10 evaluable patients per cohort will be enrolled. The maximum number of patients to be enrolled in the dose escalation and dose confirmation parts of the study combined will be 38 evaluable patients for both induction chemotherapy regimens.

For each patient, there will be a screening period of up to 21 days, a treatment period consisting of approximately 126 days (GPOH cohort) or 80 days (rapid COJEC cohort), an end of treatment visit at the end of induction treatment and a post-discontinuation safety visit 30 days after the last administration of DB. Patients will enter the follow up phase after completing the induction treatment. We recommend to follow country/site protocol/guidelines for the management of the patients after the induction treatment (e.g. High Risk-NeuroBLastoma (HR-NBL)-2 study (EudraCT : 2019-001068-31).

There are two study periods:

The first period lasts until the last patient has completed the end of treatment visit. The analysis of these results will answer the primary endpoint of the study. The planned duration for each patient enrolled is approximately 5 months, and the total study duration is approximately 2 years.

The second period lasts until the last patient has completed the follow up. In this period, data for exploratory endpoints are collected. The plan is to report late toxicity (mainly related to the high-dose chemotherapy) when the last patient completed the end of study visit and in a further report the results of 3 and 5 years follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of neuroblastoma Stage M, according to the SIOPEN modified International Neuroblastoma Risk Group (INRG) and to the INSS criteria (Appendix 1).
2. Age ≥18 months and <18 years.
3. Body weight >12 kg.
4. Alanine transaminase and aspartate aminotransferase <10 × upper limit of normal (ULN), total bilirubin <1.5 × ULN based on age specific reference ranges.
5. Calculated glomerular filtration rate > 60 mL/min/1.73 m2 or serum creatinine <1.5 × ULN corrected for age.
6. Shortening fraction (SF) ≥27% and/or left ventricular ejection fraction (LVEF) >50% as determined by echocardiography or MUGA.
7. Able to comply with scheduled follow-up and study procedures.
8. Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study specific screening procedures are conducted, according to local, regional or national law and legislation.

Exclusion Criteria:

1. Previous cancer-specific treatment for neuroblastoma.
2. Current use of a prohibited medication or requires any of these medications during the study:

   1. Treatment with corticosteroids is not allowed within 2 weeks prior to the first block of chemotherapy and until 1 week after the last treatment course with dinutuximab beta, except for life-threatening conditions.
   2. Vaccinations (including seasonal influenza) are not allowed during administration of dinutuximab beta and until 10 weeks after last treatment course.
   3. Concomitant use of intravenous (IV) immunoglobulins is not allowed.
   4. Concomitant use of cardioprotectant dexrazoxane is not allowed.
3. Pregnancy or positive pregnancy test in females of childbearing potential.
4. Breast feeding.
5. Sexually active participants not willing to use highly effective contraceptive method
6. Major surgery within 21 days prior to the first treatment dose
7. History or documented evidence of severe acute or chronic infection or infectious illness requiring parenteral therapy unless fully healed
8. Patients with spinal cord involvement
9. Any other disease, metabolic or psychological dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug
10. Have a known immediate or delayed hypersensitivity reaction to study drugs

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of dose limiting toxicities (DLTs) associated with the combination of Dinituximab Beta with GPOH chemotherapy regimen | Within first 63 days of treatment
  Number of DLT's per dose level of Dinituximab Beta
the incidence of dose limiting toxicities (DLTs) associated with the combination of Dinituximab Beta with rapid COJEC chemotherapy regimen | Within first 50 days of treatment
  Number of DLT's per dose level of Dinituximab Beta

SECONDARY OUTCOMES:
overall response rate during after Dinituximab Beta with GPOH chemotherapy regimen | 126 days
  Tumor imaging
metastatic response rate after Dinituximab Beta with GPOH chemotherapy regimen | 126 days
  Tumor imaging
overall response rate during after Dinituximab Beta with rapid COJEC chemotherapy regimen | 80 days
  Tumor imaging
metastatic response rate after Dinituximab Beta with rapid COJEC chemotherapy regimen | 80 days
  Tumor imaging

OTHER OUTCOMES:
event free survival (EFS) from the date of enrollment | 5 years
  exploratory endpoints
overall survival (OS) from the date of enrollment | 5 years
  exploratory endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Holger Lode, MD, PhD, Principal Investigator — Princess Maxima Center for Pediatric Oncology
Locations (1):
- Princess Maxima center for pediatric oncology, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication (CSR)
Supporting Information: CSR
Time Frame: Within 6 months from study end.